CLINICAL TRIAL: NCT05777356
Title: Pilot Study: Collection of Urine From Sanitary Napkins for the Analysis of Micronutrient Deficiencies
Brief Title: Sanitary Napkins for Urinary Assessment of Micronutrients
Status: Completed | Type: Observational
Sponsor: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Maren Podszun, Dr. rer. nat. Maren Podszun, University of Hohenheim
Other Study IDs: NapUrine
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Focus: Nutritional Deficiency
MeSH Terms: interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Omivorous: Healthy volunteers without dietary restrictions
  Interventions: Diagnostic Test: Urine collection and assessment of dietary intake by food frequency questionaire
- Vegetarians: Healthy volunteers who do not consume meat products
  Interventions: Diagnostic Test: Urine collection and assessment of dietary intake by food frequency questionaire
- Vegans: Healthy volunteers who do not consume any animal product
  Interventions: Diagnostic Test: Urine collection and assessment of dietary intake by food frequency questionaire

INTERVENTIONS:
Diagnostic Test: Urine collection and assessment of dietary intake by food frequency questionaire — urinary iodine, creatinine and methylmalonic acid, iodine and vitamin B12 dietary intake from foods and supplements

SUMMARY:
This study aims to find an easy urinary collection method for the assessment of urinary markers of micronutrient status.

DETAILED DESCRIPTION:
Urinary collection in newborns and infants can be difficult. Our study aims to find an easy and cheap alternative to urinary collection bags and specialized pads that can be used to measure biomarkers of iodine and vitamin B12 status in urine and can be employed in large scale trials. Using correlation analyses, the association of urinary iodine and methylmalonic acid from healthy volunteers will be assessed between untreated sample and a sample expressed from a sanitary napkin. Participants will be recruited based on their dietary pattern (omnivorous, vegetarian and vegans) to have a broad spectrum of analyte concentration. Participants weight, height, age, nutritional supplement use and diet will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers Written informed consent

Exclusion Criteria:

BMI < 18,5 and >24,9 Use of medication (except contraceptives) Smoking

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants are primarily recruited at the University of Hohenheim
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Correlation untreated and expressed urine | 8-9 weeks after completion
  Correlation of creatinine, methylmalonic acid and iodine between unprocessed urine and urine expressed from a sanitary diaper to evaluate possible matrix effects on analytes.

SECONDARY OUTCOMES:
Correlation of urinary biomarkers with food and supplement intake | 8-9 weeks after completion
  Correlation of dietary intake assessed by a food frequency questionnaire with urinary iodine and methylmalonic acid normalized to creatinine.

OTHER OUTCOMES:
Mean difference of urinary biomarkers between groups | 8-9 weeks after completion
  Exploratory analysis of differences by dietary group in urinary iodine nomalized to creatinin.
Mean difference of urinary biomarkers between groups | 8-9 weeks after completion
  Exploratory analysis of differences by dietary group in methylmalonic acid nomalized to creatinin.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No